CLINICAL TRIAL: NCT04859257
Title: Exploring the Biological Basis of Chronic Fatigue Syndrome
Acronym: CHROME
Status: Completed | Type: Observational
Sponsor: DxTerity Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: DXT-MCD-AH01
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Disease Group: Cohort 1 (Disease Group) of the study will collect blood and urine samples from participants who are either diagnosed with Chronic Fatigue Syndrome (CFS) or Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS) or experience symptoms of profound fatigue based on the cohort specific inclusion criteria.
- Control Group: Cohort 2 (Control Group) of the study will collect blood and urine samples from participants who have NOT been diagnosed with Chronic Fatigue Syndrome (CFS) or Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS) or experience symptoms of profound fatigue based on the cohort specific exclusion criteria.

SUMMARY:
To collect blood and urine samples from patients with Chronic Fatigue Syndrome (CFS), myalgic encephalomyelitis (ME), and SEID (Systemic Exertion Intolerance Syndrome) and controls for genomic, viral and metabolomic testing.

DETAILED DESCRIPTION:
To analyze gene expression (genomic) and viral analysis data from patients diagnosed with ME/CFS, the study will collect blood samples (finger stick) and information from up to 500 subjects for analysis. In addition, urine will be collected for all subjects to evaluate the study subject's metabolomics.

All participants will complete a single Study Collection event consisting of at least one MCD (2nd sample is optional) and one urine collection from home: 10% of each group (ME/CFS and Control) will complete a second Study Collection event approximately 1 to 2 weeks after the initial Study Collection. The second collection is to compare data between two collections from the same participants to observe any time-related changes in the results.

ELIGIBILITY:
Inclusion Criteria: (Cohort 1)

1. Male and female patients age 18 or older at the time of consent
2. Have a permanent address in the United States for the duration of the study
3. Have an email address and access to the internet for the duration of the study
4. Able to provide unassisted informed consent
5. Medical Record Consent (optional)
6. Diagnosed with Chronic Fatigue Syndrome (CFS) or Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS) OR
7. Report experiencing one or more of the following symptoms (record all that apply):

   1. Greatly lowered ability to perform normal daily activities due to profound fatigue that has lasted for at least 6 months
   2. Worsening of (fatigue) symptoms after physical or mental activity that would not have caused a problem before illness (post-exertional malaise).
   3. Sleep Problems. Feel overly tired or unrefreshed even after a full night of sleep
   4. Problems with thinking and memory (trouble thinking quickly, remembering things, paying attention to details, have "brain fog") OR
   5. Worsening of symptoms while standing or sitting upright -

Exclusion Criteria:

* Pregnancy

Inclusion Criteria: (Cohort 2)

1. Male and female patients age 18 or older at the time of consent
2. Have a permanent address in the United States for the duration of the study
3. Have an email address and access to the internet for the duration of the study
4. Able to provide unassisted informed consent
5. Medical Record Consent (optional)

Exclusion Criteria:

1. Pregnant
2. Diagnosed with Chronic Fatigue Syndrome (CFS) or Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS) OR
3. Report experiencing one or more of the following symptoms (record all that apply):

   1. Greatly lowered ability to perform normal daily activities due to profound fatigue that has lasted for at least 6 months
   2. Worsening of (fatigue) symptoms after physical or mental activity that would not have caused a problem before illness (post-exertional malaise).
   3. Sleep Problems. Feel overly tired or unrefreshed even after a full night of sleep
   4. Problems with thinking and memory (trouble thinking quickly, remembering things, paying attention to details, have "brain fog") OR
   5. Worsening of symptoms while standing or sitting upright

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1 of this study will collect blood sample and a urine sample from up to 150 subjects who are either diagnosed with CFS/ME or experience symptoms of fatigue.
  Cohort 2 (Control Group) of the study will collect blood and urine samples from participants who have NOT been diagnosed with Chronic Fatigue Syndrome (CFS) or Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS) or experience symptoms of profound fatigue based on the cohort specific exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Collect blood samples from patients with Chronic Fatigue Syndrome (CFS), myalgic encephalomyelitis (ME), and Systemic Exertion Intolerance Syndrome (SEID), and controls for genomic testing. | 3 months
  To enable research focused on discriminating differentiated symptoms of various sources of CFS from other autoimmune and viral pathogenesis of disease which could prove valuable in researching for inflammation and immunity related therapeutics.
Collect blood samples from patients with Chronic Fatigue Syndrome (CFS), myalgic encephalomyelitis (ME), and Systemic Exertion Intolerance Syndrome (SEID), and controls for viral testing. | 3 months
  To enable research focused on discriminating differentiated symptoms of various sources of CFS from other autoimmune and viral pathogenesis of disease which could prove valuable in researching for inflammation and immunity related therapeutics.
Collect urine samples from patients with Chronic Fatigue Syndrome (CFS), myalgic encephalomyelitis (ME), and Systemic Exertion Intolerance Syndrome (SEID), and controls for metabolomic testing. | 3 months
  To enable research focused on discriminating differentiated symptoms of various sources of CFS from other autoimmune and viral pathogenesis of disease which could prove valuable in researching for inflammation and immunity related therapeutics.

CONTACTS AND LOCATIONS:
Locations (1):
- DxTerity Diagnostics Inc., Compton, California, United States